CLINICAL TRIAL: NCT01793688
Title: Special Use-result Surveillance Of Unasyn-s (Kit) For Intravenous Use - A Surveillance On High-dose (>6 G Daily) Administration For Pneumonia, Lung Abscess And Peritonitis -
Brief Title: Special Use-Result Surveillance of Unasyn-S (Kit) for Intravenous Use - A Surveillance on High-dose (>6 g Daily) Administration -
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A9231002
Record Dates: First submitted 2013-02-04; First posted 2013-02-15 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Pneumonia; Lung Abscess; Peritonitis
Keywords: UNASYN-S; High Dose
MeSH Terms: conditions — Pneumonia; Lung Abscess; Peritonitis | interventions — Sulbactam; Ampicillin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sulbactam Sodium/Ampicillin Sodium: Patients with the following disease who received high doses of UNASYN (exceeding 6 g per day) by intravenous injection or intravenous drip infusion from the first dosing date or the second dosing date: Pneumonia, Lung Abscess, Peritonitis.
  Interventions: Drug: Sulbactam Sodium/Ampicillin Sodium

INTERVENTIONS:
Drug: Sulbactam Sodium/Ampicillin Sodium — Intravenous use; The usual adult dosage is 6 g of sulbactam sodium and ampicillin sodium (potency) per day given in two divided doses via intravenous injection or drip infusion. In the case of severe infection, the dosage may be increased if appropriate. Maximum dosage should not exceed 3 g (potency) 4 times daily (daily dose of 12 g (potency)).
  Kit for intravenous use; The usual adult dosage is 6 g of sulbactam sodium and ampicillin sodium (potency) per day given in two divided doses via intravenous injection after dissolved in an accompanying reconstitution diluent. In the case of severe infection, the dosage may be increased if appropriate. Maximum dosage should not exceed 3 g (potency) 4 times daily (daily dose of 12 g (potency)).
  Other Names: UNASYN-S

SUMMARY:
The purpose of the survey is to study the followings under practical use, regarding the safety and effectiveness in high-dose administration (exceeding 6 g per day) of UNASYN-S and UNASYN-S KIT for intravenous use (UNASYN).

1. Adverse Drug Reaction(s) that cannot be expected from precautions (Unexpected Adverse Drug Reaction)
2. Incidence status of adverse drug reactions
3. Factors that may affect the safety and effectiveness

DETAILED DESCRIPTION:
Implemented as a Special Investigation by a central registration system. Secondary data collection. Safety and effectiveness of UNASYN-S under Japanese medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following disease who received high doses of UNASYN (exceeding 6 g per day) from the first dosing date or the second dosing date. 1) Pneumonia, 2) Lung Abscess, 3) Peritonitis
* Patients aged 15 years or more

Exclusion Criteria:

* Patients with the following disease who received high doses of UNASYN (less than 6 g per day) from the first dosing date or the second dosing date. 1) Pneumonia, 2) Lung Abscess, 3) Peritonitis
* Patients aged less than 15 years.

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with the following disease who received high doses of UNASYN (exceeding 6 g per day) from the first dosing date or the second dosing date.
  1. Pneumonia
  2. Lung Abscess
  3. Peritonitis
Sampling Method: Probability Sample
Enrollment: 982 (Actual)
Dates: Start 2013-03-12 (Actual); Primary Completion 2016-01-27 (Actual); Study Completion 2016-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9231002&StudyName=Drug%20Use%20Investigation%20Of%20Sulbactam/Ampicillin%20%28UNASYN%29%2012g%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total 986 subjects were registered in this study. Of the 986 subjects, 982 subjects CRFs were collected and included in the study.Of the 982 subjects, 2 subjects were excluded from the safety analysis set (SAS). In total, 980 subjects were included in the SAS as the completed the study.
Groups:
- Sulbactam Sodium/Ampicillin Sodium: The usual adult dosage was 6 g daily (strength) in two divided doses as sulbactam sodium/ampicillin sodium given by intravenous injection or intravenous drip infusion. In cases of severe infection, the dose could be increased with a maximum dose of 3 g (strength) four times daily (12 g [strength] daily).
Period: Overall Study
Arm/Group | Sulbactam Sodium/Ampicillin Sodium
Started | 982
Completed | 980
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: A total 986 subjects were registered in this study. Of the 986 subjects, 982 subjects CRFs were collected and included in the study.Of the 982 participants, 2 participants were excluded from the baseline analysis due to a protocol violation.
Arm/Group | Sulbactam Sodium/Ampicillin Sodium
Number analyzed (Participants) | 980
Age, Customized [Number; unit: Participants]
  >=15 and <65 years | 255
  ˃=65 years | 725
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 296
  Male | 684
Diagnosis [Number; unit: Participants]
  Pneumonia | 861
  Lung Abscess | 71
  Peritonitis | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sulbactam sodium/ampicillin sodium in a participant who received sulbactam sodium/ampicillin sodium. Relatedness to sulbactam sodium/ampicillin sodium was assessed by the investigator.
Time Frame: 14 Days
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria of the study, and who had been received sulbactam sodium/ampicillin sodium at least once.
Measure: Number; unit: Participants
Arm/Group | Sulbactam Sodium/Ampicillin Sodium
Number analyzed (Participants) | 980
Participants | 96

2. Primary Outcome: Clinical Effectiveness Rate by Indication
Description: Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of participants with assessable effectiveness evaluation, was presented by each indication (pneumonia, lung abcess and peritorinitis) along with the corresponding exact 2-sided 95% confidence interval. Overall effectiveness of sulbactam sodium/ampicillin sodium was determined by the investigator based on clinical symptoms and examinations at the end of high-dose (>6 g daily) treatment. Clinical effectiveness was assessed according to the following categories: (1) effective, (2) ineffective, or (3) unassessable at the end of treatment.
Time Frame: 14 Days
Population: The effectiveness analysis set comprised of participants in safety analysis set who had effectiveness evaluation at least once.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sulbactam Sodium/Ampicillin Sodium
Number analyzed (Participants) | 978
Percentage of participants
  With Pneumonia (n=856) | 85.1 [82.4 to 87.5]
  With Lung Abcess (n=70) | 78.5 [66.5 to 87.7]
  With Peritonitis (n=47) | 78.7 [64.3 to 89.3]

3. Secondary Outcome: Number of Participants With Treatment-Related Serious Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sulbactam sodium/ampicillin sodium in a participant who received sulbactam sodium/ampicillin sodium. A treatment-related serious adverse event was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Relatedness to sulbactam sodium/ampicillin sodium was assessed by the investigator.
Time Frame: 14 Days
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sulbactam Sodium/Ampicillin Sodium
Number analyzed (Participants) | 980
Participants | 6

4. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events Unexpected From Japanese Package Insert
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sulbactam sodium/ampicillin sodium in a participant who received sulbactam sodium/ampicillin sodium. Expectedness of the adverse event was determined according to Japanese package insert. Relatedness to sulbactam sodium/ampicillin sodium was assessed by the investigator.
Time Frame: 14 Days
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sulbactam Sodium/Ampicillin Sodium
Number analyzed (Participants) | 980
Participants | 30

ADVERSE EVENTS:
Arm/Group | Sulbactam Sodium/Ampicillin Sodium
Serious Adverse Events (participants affected / at risk) | 43/980
Other Adverse Events (participants affected / at risk) | 158/980
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sulbactam Sodium/Ampicillin Sodium (N=980)
Infectious pleural effusion (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Lung infection (Infections and infestations) | 2
Lung abscess (Infections and infestations) | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2
Adrenal disorder (Endocrine disorders) | 1
Marasmus (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Hemiplegia (Nervous system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3
Gastric ulcer (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Disease progression (General disorders) | 2
Multi-organ failure (General disorders) | 1
White blood cell count increased (Investigations) | 1
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.50% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sulbactam Sodium/Ampicillin Sodium (N=980)
Decreased appetite (Metabolism and nutrition disorders) | 9
Anaemia (Blood and lymphatic system disorders) | 8
Aspartate aminotransferase increased (Investigations) | 8
Pyrexia (General disorders) | 7
Restlessness (Psychiatric disorders) | 6
Delirium (Psychiatric disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6
Liver disorder (Hepatobiliary disorders) | 6
Alanine aminotransferase increased (Investigations) | 6
Diarrhoea (Gastrointestinal disorders) | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Hypokalaemia (Metabolism and nutrition disorders) | 12
Insomnia (Psychiatric disorders) | 11
Hepatic function abnormal (Hepatobiliary disorders) | 11
Constipation (Gastrointestinal disorders) | 10
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Protein total decreased (Investigations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.